CLINICAL TRIAL: NCT05017480
Title: A Double-blind, Multi-center, Randomized Controlled Clinical Study to Evaluate the Efficacy and Safety of CBP-201 in Chinese Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Evaluate the Efficacy and Safety of CBP-201 in Moderate to Severe Atopic Dermatitis in China
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Connect Biopharm LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBP-201-CN002
Record Dates: First submitted 2021-08-13; First posted 2021-08-23 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Moderate-to-severe Atopic Dermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBP-201 Dose (Experimental): CBP-201 Dose subcutaneous (SC) injection
  Interventions: Drug: CBP-201
- Placebo (Placebo Comparator): subcutaneous (SC) injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CBP-201 — CBP-201 subcutaneous(SC) injection.
  Arms: CBP-201 Dose
Drug: Placebo — subcutaneous(SC) injection
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of CBP-201 in Chinese subjects with moderate to severe atopic dermatitis.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, multi-center, controlled study designed to assess the efficacy, safety and PK characteristics of CBP-201 in eligible subjects with moderate to severe AD.

The study includes a screening period, a treatment period and a follow-up period. The treatment period is divided into two stages.

ELIGIBILITY:
Inclusion Criteria:

1. 12≤ age ≤75 years at the screening visit, male or female;
2. Diagnosed with atopic dermatitis (according to the American Academy of Dermatology's Guidelines of care for the management of atopic dermatitis, 2014[1]) at the screening, visit and:

   a) The subject has been suffering from the disease for more than 1 year at the time of screening, and according to the judgment of the investigator, the subject has had poor response to topical drugs such as corticosteroids, phosphodiesterase-4 (PDE-4) inhibitors or calcineurin inhibitors (TCI), or it is not medically suitable for the subject to receive topical drug treatment (e.g., there are important side effects or safety risks);

   Note: Poor response is defined as any of the following conditions:

   i. The patient has not achieved and maintained response or reached a low disease activity state (equivalent to IGA 0=asymptomatic to 2=mild) despite regular use of topical therapy during the 1 year before baseline; ii. The patient has received systemic treatment for AD despite regular use of topical therapy during the 1 year before baseline.

   b. At the screening and baseline visit, Investigator's Global Assessment (IGA) score ≥3 (according to the validated Investigator Global Assessment for Atopic Dermatitis [vIGA-AD™] scale, see Section 17.4 Appendix D), Eczema Area and Severity Index (EASI) score≥16 (see Section 17.5, Appendix E), and≥10% body surface area (BSA) of AD involvement(see Section 17.6, Appendix F); c. The average score of the maximum pruritus intensity in the Peak Pruritus Numerical Rating Scale (PP-NRS) ≥4 (see Section 17.1, Appendix A).

   Note: The baseline average score of maximum pruritus intensity in the PP-NRS will be calculated based on the average value of the maximum pruritus intensity in the PP-NRS score [daily score range 0-10] every day within 7 days before randomization. In these 7 days, the scores of at least 4 days are required for the calculation of the baseline average score. If the patient's reporting days are less than 4 days in the 7 days before the planned date of randomization, randomization should be postponed until the requirements are met, but it is not allowed to exceed the maximum screening period of 28 days.
3. Able and willing to use a stable dose of a mild emollient at the AD involvement area twice a day starting from at least 7 days before baseline and continue to use it during the study period (see Section 8.1.1.2 Emollients).
4. Female subjects of childbearing potential (FCBP) and male subjects who have not undergone vasectomy must take highly effective contraceptive measures during the entire study period, including the 8-week follow-up period after discontinuation of study drug. Postmenopausal women (determined by testing follicle stimulating hormone [FSH]) and women with a record of surgical sterilization (i.e., tubal ligation or hysterectomy or bilateral oophorectomy) before the screening visit can be considered infertile.

   Highly effective contraceptive measures include:

   i. Abstinence (acceptable only if it is part of the subject's routine lifestyle); ii. Hormones (oral, patch, ring, injection, implant) combined with male condoms. This measure must be used at least 30 days before the first study drug administration. Otherwise, another acceptable method of contraception must be used; iii. Intrauterine device (IUD) combined with male condoms; iv. Exceptions are: a) women who have had amenorrhea for at least 12 consecutive months without using drugs known to cause amenorrhea, and have a recorded FSH level greater than 40 mIU/mL or in the postmenopausal range; or b) surgical sterilization (e.g., hysterectomy, bilateral oophorectomy).
5. Subjects and/or their guardians have the ability to learn the study requirements and process, and voluntarily take part in the clinical trial and sign an informed consent form (ICF); note: for subjects ≥18 years: subjects voluntarily agree to take part in the study by themselves and sign ICF; for subjects aged 12-17 years: subjects and their guardians voluntarily agree to take part in the study, the guardians sign the ICF, and the subjects sign the informed assent form for minors by themselves.
6. Subjects and/or their guardians are willing and able to comply with study visits and related procedures.

Exclusion Criteria:

1. Patients who have received any of the following treatments:

   1. Treatment with dupilumab or any anti-IL-4Rα or IL-13 antibodies;
   2. Topical drugs for treatment of AD or have the potential to affect the assessment of AD, including but not limited to corticosteroids, PDE-4 inhibitors, Janus kinase (JAK) inhibitors, aromatic hydrocarbon receptor agonists, tacrolimus or pimecrolimus, or traditional Chinese medicine (TCM) or herbal medicine, etc. within 2 weeks before baseline;
   3. Have undergone bleaching baths ≥ twice within 2 weeks before baseline;
   4. Have begun to use prescription emollients or emollients containing additives (e.g., ceramide, hyaluronic acid, urea, or filaggrin breakdown products) to treat AD from the screening period (if the subject has started using this kind of emollient before the screening visit, they can continue to use it at a stable dose; if the subject is intolerable to the emollients provided uniformly by the sponsor during the screeing period, he/she can change to emollient of this kind used previously, but it must be used at a stable dose for at least 7 days before baseline and during the study period);
   5. Treatment with systemic corticosteroids or other immunosuppressive/immunomodulating substances (e.g., cyclosporine, mycophenolate mofetil, azathioprine, methotrexate, or oral JAK inhibitors) due to AD or other diseases within 4 weeks before baseline (except for corticosteroid inhalers and nasal sprays);
   6. Treatment with systemic TCM or herbal treatment within 4 weeks before baseline (note: except for those for the treatment of diseases other than AD, which are necessary and will neither increase the risks of the subjects nor affect the assessment of the study in accordance with the medical judgements of the investigator and/or specialist physician);
   7. Treatment with phototherapy (narrow band ultraviolet B [NBUVB], ultraviolet B [UVB], ultraviolet A1 [UVA1], psoralen + ultraviolet A [PUVA]), sunbed or any other light emitting device (LED) therapy within 4 weeks before baseline;
   8. Have used any investigational drug/treatment within 4 weeks before baseline or 5 drug half-lives, whichever is longer;
   9. Treatment with other biological agents (e.g., omalizumab) within 3 months before baseline or 5 drug half-lives (if known), whichever is longer;
   10. Have been vaccinated with live (attenuated) vaccine within 8 weeks before baseline;
   11. Treatment with cell depletion agents (e.g., rituximab) within 6 months before baseline;
   12. Treatment with allergen specific immunotherapy (SIT) within 6 months before baseline (except those who were already on stable-dose therapy before baseline).

   Eligibility criteria Inclusion criteria

   Patients must meet all of the following criterias to be enrolled into this study:
2. Patients who meet any of the following:

   1. History of hypersensitivity to L-histidine, trehalose or Tween 80;
   2. Other skin complications in addition to AD that may interfere with the study assessments;
   3. Any history of vernal keratoconjunctivitis (VKC) and atopic keratoconjunctivitis (AKC);
   4. History of malignant tumor within 5 years before screening, except for cervical carcinoma in situ or non-metastatic cutaneous squamous cell carcinoma or basal cell carcinoma;
   5. Active tuberculosis (TB) at the screening visit, latent tuberculosis or a history of non-tuberculous Mycobacterium infection

   Note:
   * Unless there is a clear specialist record proving that the patient has received adequate treatment and is currently able to start receiving biological treatment (based on the medical judgment of the investigator and/or infectious disease specialist);
   * If necessary, T-spot test may be used for auxiliary diagnosis of suspected tuberculosis patients; f. Positive for hepatitis B surface antigen (HBsAg), or positive for hepatitis B core antibody (HBcAb) and HBV-DNA, or positive for hepatitis C antibody and HCV RNA polymerase chain reaction; or serologically positive for human immunodeficiency virus (HIV) at the screening visit; g. Any of the following laboratory test abnormalities at the screening visit: i. Aspartate aminotransferase or alanine aminotransferase > 2 times the upper limit of normal (ULN), or total bilirubin > 1.5×ULN ii. Serum creatinine > 1.2×ULN iii. Hemoglobin < 8.5 g/dl (85.0 g/L) in male patients and < 8.0 g/dl (80.0 g/L) in female patients iv. White blood cell count <3.0×109/L or ≥14×109/L v. Platelet count <100×109/L h. Planning to undergo major surgical operations during the study period; i. Used systemic treatment with antibiotics, antiviral drugs, antiparasitic drugs, antigenic drugs, or antifungal drugs due to infection within 4 weeks before the baseline visit, or suffered from superficial skin infection (e.g., impetigo) within 2 weeks before baseline (after the infection subsides, the subjects can be rescreened); j. History of parasite infection (e.g., helminth) within 6 months before baseline; k. According to the investigator's judgment, there is a known or suspected history of immunosuppression within 6 months before baseline, including a history of invasive opportunistic infections, such as aspergillosis, coccidiosis, histoplasmosis, HIV, listeriosis, Pneumocystis or tuberculosis, even if the infection has subsided; or there is an abnormally frequently recurrent or persistent infection; l. History of alcohol or drug abuse within 2 years before the screening visit; m. Any other medical or psychological condition (including clinically significant laboratory test abnormalities, ECG parameters, etc.) at the screening visit, which, as judged by the investigator, may indicate new and/or insufficiently understood diseases, may put the patient at an unreasonable risk due to his/her participation in the clinical trial, may lead to unreliable results of the patient's participation, or may interfere with the study assessments. The specific reasons for patients excluded due to this criterion will be indicated in the study documents (medical records, eCRF, etc.).
3. Pregnant or lactating women, or subjects with pregnancy or lactation plans during the study period.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzhou Connect, Study Director — Connect Biopharm LLC
Locations (48):
- China (48):
  - Connect Investigative Site 33, Hefei, Anhui
  - Connect Investigative Site 01, Beijing, Beijing Municipality
  - Connect Investigative Site 02, Beijing, Beijing Municipality
  - Connect Investigative Site 03, Beijing, Beijing Municipality
  - Connect Investigative Site 17, Beijing, Beijing Municipality
  - Connect Investigative Site 47, Beijing, Beijing Municipality
  - Connect Investigative Site 28, Chongqing, Chongqing Municipality
  - Connect Investigative Site 29, Chongqing, Chongqing Municipality
  - Connect Investigative Site 30, Chongqing, Chongqing Municipality
  - Connect Investigative Site 36, Chongqing, Chongqing Municipality
  - Connect Investigative Site 38, Fuzhou, Fujian
  - Connect Investigative Site 07, Guangzhou, Guangdong
  - Connect Investigative Site 25, Guangzhou, Guangdong
  - Connect Investigative Site 37, Guangzhou, Guangdong
  - Connect Investigative Site 46, Guangzhou, Guangdong
  - Connect Investigative Site 48, Guangzhou, Guangdong
  - Connect Investigative Site 43, Shaoguan, Guangdong
  - Connect Investigative Site 52, Shenzhen, Guangdong
  - Connect Investigative Site 41, Haikou, Hainan
  - Connect Investigative Site 42, Haikou, Hainan
  - Connect Investigative Site 20, Zhengzhou, He'an
  - Connect Investigative Site 32, Shijiazhuang, Hebei
  - Connect Investigative Site 45, Nanyang, Henan
  - Connect Investigative Site 54, Xinxiang, Henan
  - Connect Investigative Site 49, Wuhan, Hubei
  - Connect Investigative Site 35, Baotou, Inner Mongolia
  - Connect Investigative Site 26, Nanjing, Jiangsu
  - Connect Investigative Site 18, Suzhou, Jiangsu
  - Connect Investigative Site 55, Wuxi, Jiangsu
  - Connect Investigative Site 10, Zhenjiang, Jiangsu
  - Connect Investigative Site 34, Nanchang, Jiangxi
  - Connect Investigative Site 44, Yinchuan, Ningxia
  - Connect Investigative Site 11, Jinan, Shandong
  - Connect Investigative Site 50, Jinan, Shandong
  - Connect Investigative Site 51, Jinan, Shandong
  - Connect Investigative Site 12, Yantai, Shandong
  - Connect Investigative Site 08, Taiyuan, Shanxi
  - Connect Investigative Site 24, Taiyuan, Shanxi
  - Connect Investigative Site 39, Yuncheng, Shanxi
  - Connect Investigative Site 05, Tianjin, Tianjin Municipality
  - Connect Investigative Site 06, Tianjin, Tianjin Municipality
  - Connect Investigative Site 13, Shanxi, Xi'an
  - Connect Investigative Site 22, Ürümqi, Xinjiang
  - Connect Investigative Site 53, Qujing, Yunnan
  - Connect Investigative Site 14, Hangzhou, Zhejiang
  - Connect Investigative Site 15, Hangzhou, Zhejiang
  - Connect Investigative Site 16, Hangzhou, Zhejiang
  - Connect Investigative Site 19, Jinhua, Zhejiang

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: CBP-201 300mg Q2W: The subjects receive a subcutaneous injection of CBP-201 600 mg on Day 1, begin to receive a subcutaneous injection of CBP-201 300 mg (2 ml) from Week 2 (W2), and receive treatment at the same dose every 2 weeks thereafter(Q2W) until W14.
- Group B: Placebo Q2W: The subjects receive a subcutaneous injection of placebo 4 ml, begin to receive a subcutaneous injection of placebo 2 ml from W2, and receive placebo 2 ml every 2 weeks (Q2W) thereafter until W14.
- Group C: Double-blinded CBP-201 300mg Q2W: Subjects who have achieved EASI-50 in the W16 pre-administration treatment assessment will be 1:1 randomized to one of the following two groups to receive study treatment starting from W16:
  The subjects receive a subcutaneous injection of CBP-201 300 mg every 2 weeks (Q2W) until W50.
- Group D: Double-blinded CBP-201 300mg Q4W: Subjects who have achieved EASI-50 in the W16 pre-administration treatment assessment will be 1:1 randomized to one of the following two groups to receive study treatment starting from W16:
  The subjects receive a subcutaneous injection of CBP-201 300 mg every 4 weeks. In order to maintain the injection every 2 weeks blind, when not receiving CBP-201, the subjects receive an injection of placebo 2 ml once every 4 weeks until W50.
- Group E: Open-Label CBP-201 300mg Q2W: Subjects who have not achieved EASI-50 in the W16 pre-administration treatment assessment will receive the following treatment starting from W16:
  The subjects receive a subcutaneous injection of CBP-201 300 mg every 2 weeks until W50.
Period: Stage 1 Study
Arm/Group | Group A: CBP-201 300mg Q2W | Group B: Placebo Q2W | Group C: Double-blinded CBP-201 300mg Q2W | Group D: Double-blinded CBP-201 300mg Q4W | Group E: Open-Label CBP-201 300mg Q2W
Started | 219 | 111 | 0 | 0 | 0
Completed | 209 | 102 | 0 | 0 | 0
Not Completed | 10 | 9 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 6 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0
Not completed — Poor Compliance | 1 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0
Period: Stage 2 Study
Arm/Group | Group A: CBP-201 300mg Q2W | Group B: Placebo Q2W | Group C: Double-blinded CBP-201 300mg Q2W | Group D: Double-blinded CBP-201 300mg Q4W | Group E: Open-Label CBP-201 300mg Q2W
Started | 0 | 0 | 113 | 112 | 86
Completed | 0 | 0 | 107 | 99 | 73
Not Completed | 0 | 0 | 6 | 13 | 13
Not completed — Withdrawal by Subject | 0 | 0 | 6 | 9 | 11
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0
Not completed — COVID-19 | 0 | 0 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: CBP-201 300mg Q2W | Group B: Placebo Q2W | Total
Number analyzed (Participants) | 219 | 111 | 330
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (16.65) | 39.6 (17.54) | 38.9 (16.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 40 | 113
  Male | 146 | 71 | 217
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 219 | 111 | 330
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 23.66 (3.932) | 24.98 (4.829) | 24.10 (4.293)
Severity of Atopic Dermatitis at Baseline [Count of Participants; unit: Participants] — IGA: Validated Investigator Global Assessment
  The Validated Investigator Global Assessment for AD (vIGA-AD™) Scale is a 5-point classification scale based on the overall appearance of the skin lesions at a specific time point (0=clear; 1=almost clear; 2=mild; 3=moderate; 4=severe).
  Participants
    Moderate (IGA=3) | 99 | 50 | 149
    Severe (IGA=4) | 120 | 61 | 181
EASI at Baseline [Mean (Standard Deviation); unit: units on a scale] — Eczema Area and Severity Index (EASI)
  The EASI score quantifies the severity and extent of AD, as well as the severity of erythema, infiltration, excoriation and lichenification of the four anatomical regions-head and neck, trunk, upper extremities and lower extremities. The total EASI score ranges from 0 (lowest) to 72 (highest); the higher the score, the higher the severity of AD (more severe).
  units on a scale | 29.27 (11.658) | 28.62 (12.092) | 29.05 (11.791)
PP-NRS at Baseline [Mean (Standard Deviation); unit: units on a scale] — Peak Pruritus Numerical Rating Scale (PP-NRS)
  It is a single self-reported item designed to measure the peak pruritus or"worst" pruritus in the past 24 hours. The score ranges from 0 to 10, in which 0 represents "no pruritus" and 10 "worst imaginable pruritus".
  units on a scale | 7.19 (1.680) | 7.17 (1.459) | 7.18 (1.607)
BSA at Baseline [Mean (Standard Deviation); unit: units on a scale] — Percentage of body surface area (BSA) affected by AD
  The "Rule of Nines" is used to estimate the maximum percentage in each area:
  * Head and neck [9%]
  * Anterior trunk [18%]
  * Back [18%]
  * Upper limbs [18%]
  * Lower limbs [36%]
  * Genitals [1%])
  Regardless of the age of the subject, the area of the subject's entire palm (five fingers adducted together) is about 1% of the subject's BSA. As part of the EASI assessment, the number of palms in different body parts is assessed to calculate the percentage of BSA affected by AD.
  units on a scale | 48.55 (20.666) | 46.64 (21.581) | 47.91 (20.965)
SCORAD at Baseline [Mean (Standard Deviation); unit: units on a scale] — Scoring Atopic Dermatitis Index
  A clinical tool used to assess the severity of AD (extent/severity) and subjective signs/symptoms (e.g., itch/sleeplessness). The severity is determined by grading the severity of the 6 signs on a 0-3 subscale. A visual analog scale (VAS) is used to score subjective symptoms, with 0=no itch (or sleeplessness) and 10=most severe itch (or sleeplessness). The total score is the sum of extensiveness/5+7 x severity/2+VAS (symptoms). SCORAD results range from 0 and 103. The higher the score, the more severe the AD.
  units on a scale | 68 (12.940) | 67.37 (12.531) | 67.79 (12.788)
POEM at Baseline [Mean (Standard Deviation); unit: units on a scale] — Patient Oriented Eczema Measure
  It is a questionnaire composed of 7 items to assess disease symptoms on a scale of 0-4 (dryness, itching, flaking off, cracking, sleeplessness, bleeding and weeping or oozing); the scores range from 0 (no disease) to 28 (severe disease); the higher the score, the worse the quality of life.
  units on a scale | 21.4 (6.10) | 21.1 (6.13) | 21.3 (6.11)
DLQI at Baseline [Mean (Standard Deviation); unit: units on a scale] — Dermatology Life Quality Index
  It is a questionnaire containing 10 items to assess the impact of AD on quality of life (QOL) in the past week, and the scores range from 0 (no disease) to 30 (severe disease); the higher the score, the worse the quality of life. Population: Missing Data
  units on a scale
    number analyzed (Participants) | 217 | 108 | 325
    (all) | 16.0 (7.32) | 15.7 (6.11) | 15.9 (6.93)

OUTCOME MEASURES:

1. Primary Outcome: Investigator Global Assessment (IGA) (0-1)
Description: The percentage of subjects whose IGA score is 0-1 and decreased by ≥2 points
  The Validated Investigator Global Assessment for AD (vIGA-AD™) Scale is a 5-point classification scale based on the overall appearance of the skin lesions at a specific time point (0=clear; 1=almost clear; 2=mild; 3=moderate; 4=severe).
Time Frame: Baseline to Week16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: CBP-201 300mg Q2W | Group B: Placebo Q2W
Number analyzed (Participants) | 219 | 111
percentage of participants | 29.0 [23.0 to 35.0] | 5.9 [1.4 to 10.4]

2. Secondary Outcome: Eczema Area and Severity Index (EASI)-75
Description: The percentage of subjects achieving EASI-75 (EASI score is decreased by ≥75% from baseline)
  The total EASI score ranges from 0 (lowest) to 72 (highest); the higher the score, the higher the severity of AD (more severe).
Time Frame: Baseline to Week16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: CBP-201 300mg Q2W | Group B: Placebo Q2W
Number analyzed (Participants) | 219 | 111
percentage of participants | 58.6 [51.9 to 65.3] | 22.6 [14.5 to 30.7]

3. Secondary Outcome: Change in Peak Pruritus Numerical Rating Scale(PP-NRS) (Decreased by ≥ 4 Points)
Description: The percentage of subjects whose weekly average PP-NRS is decreased by ≥ 4 points
  The score ranges from 0 to 10, in which 0 represents "no pruritus" and 10 "worst imaginable pruritus".
Time Frame: Baseline to Week16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: CBP-201 300mg Q2W | Group B: Placebo Q2W
Number analyzed (Participants) | 216 | 110
percentage of participants | 36.3 [29.7 to 42.8] | 10.5 [4.5 to 16.5]

4. Secondary Outcome: Change in Peak Pruritus Numerical Rating Scale(PP-NRS) (Decreased by ≥ 3 Points)
Description: The percentage of subjects whose weekly average PP-NRS is decreased by ≥ 3 points
  The score ranges from 0 to 10, in which 0 represents "no pruritus" and 10 "worst imaginable pruritus".
Time Frame: Baseline to Week16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: CBP-201 300mg Q2W | Group B: Placebo Q2W
Number analyzed (Participants) | 218 | 111
percentage of participants | 50.0 [43.2 to 56.9] | 20.3 [12.7 to 28.0]

5. Secondary Outcome: Change in the Weekly Average Peak Pruritus Numerical Rating Scale(PP-NRS)
Description: Change in the weekly average PP-NRS
  The score ranges from 0 to 10, in which 0 represents "no pruritus" and 10 "worst imaginable pruritus".
Time Frame: Baseline to Week16
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group A: CBP-201 300mg Q2W | Group B: Placebo Q2W
Number analyzed (Participants) | 219 | 111
score on a scale | -2.95 [-3.28 to -2.62] | -0.99 [-1.46 to -0.53]

6. Secondary Outcome: Eczema Area and Severity Index (EASI)-90
Description: The percentage of subjects achieving EASI-90 (EASI score is decreased by ≥90% from baseline)
  The total EASI score ranges from 0 (lowest) to 72 (highest); the higher the score, the higher the severity of AD (more severe).
Time Frame: Baseline to Week16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: CBP-201 300mg Q2W | Group B: Placebo Q2W
Number analyzed (Participants) | 219 | 111
percentage of participants | 33.4 [27.0 to 39.8] | 6.4 [1.4 to 11.4]

7. Secondary Outcome: Percentage Change in the Weekly Average Peak Pruritus Numerical Rating Scale(PP-NRS)
Description: Percentage change in the weekly average PP-NRS
  The score ranges from 0 to 10, in which 0 represents "no pruritus" and 10 "worst imaginable pruritus".
Time Frame: Baseline to Week16
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage change of PP-NRS value
Arm/Group | Group A: CBP-201 300mg Q2W | Group B: Placebo Q2W
Number analyzed (Participants) | 219 | 111
percentage change of PP-NRS value | -40.00 [-44.80 to -35.20] | -13.50 [-20.19 to -6.82]

ADVERSE EVENTS:
Time Frame: Stage 1 treatment period (Day1~Week16) - Stage 2 treatment period (Week16~Week52) - Follow-up period (Week53~Week60)
Arm/Group | Group A: CBP-201 300mg Q2W | Group B: Placebo Q2W | Group C: Double-blinded CBP-201 300mg Q2W | Group D: Double-blinded CBP-201 300mg Q4W | Group E: Open-Label CBP-201 300mg Q2W
All-Cause Mortality (participants affected / at risk) | 0/219 | 0/111 | 0/113 | 0/112 | 0/85
Serious Adverse Events (participants affected / at risk) | 1/219 | 3/111 | 1/113 | 3/112 | 6/85
Other Adverse Events (participants affected / at risk) | 80/219 | 34/111 | 70/113 | 67/112 | 53/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: CBP-201 300mg Q2W (N=219) | Group B: Placebo Q2W (N=111) | Group C: Double-blinded CBP-201 300mg Q2W (N=113) | Group D: Double-blinded CBP-201 300mg Q4W (N=112) | Group E: Open-Label CBP-201 300mg Q2W (N=85)
Injury,poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Cardiac disorders (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Endocrine disorders (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular disorders (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorders (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: CBP-201 300mg Q2W (N=219) | Group B: Placebo Q2W (N=111) | Group C: Double-blinded CBP-201 300mg Q2W (N=113) | Group D: Double-blinded CBP-201 300mg Q4W (N=112) | Group E: Open-Label CBP-201 300mg Q2W (N=85)
Hyperlipidaemia (Metabolism and nutrition disorders) | 23 (25) | 6 (6) | 3 (3) | 8 (10) | 5 (6)
hyperuricemia (Metabolism and nutrition disorders) | 21 (22) | 5 (6) | 7 (8) | 3 (3) | 3 (3)
Atopic Dermatitis (Skin and subcutaneous tissue disorders) | 23 (31) | 19 (23) | 14 (16) | 27 (35) | 14 (20)
upper respiratory infection (Infections and infestations) | 14 (14) | 7 (7) | 12 (13) | 12 (13) | 15 (15)
Injection site erythema (General disorders) | 11 (20) | 1 (1) | 3 (4) | 6 (7) | 3 (4)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 38 (38) | 34 (35) | 21 (21)
Fever (General disorders) | 0 (0) | 0 (0) | 9 (10) | 9 (9) | 7 (8)
urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (6) | 6 (7) | 5 (6)
Tested positive for SARS-CoV-2 (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 7 (7) | 2 (2)
conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 3 (5) | 6 (6)
Elevated alanine aminotransferase (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 5 (5)
Weight Gain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 6 (8) | 1 (1) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT05017480/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT05017480/SAP_001.pdf